CLINICAL TRIAL: NCT06642714
Title: Early Non-invasive Ventilation and Progressive High Flow Oxygen Therapy Through Tracheostomy Tube Weaning Protocol in Tracheostomized Patients with Prolonged Mechanical Ventilation: a Prospective Cohort Study
Brief Title: Early Non-invasive Ventilation and Progressive High Flow Oxygen Therapy Through Tracheostomy Tube Weaning Protocol in Tracheostomized Patients with Prolonged Mechanical Ventilation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jingyi Ge, Principal Investigator, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018Z-001
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mechanical Ventilation; Weaning from Mechanical Ventilation
Keywords: tracheostomy; mechanical ventilation; non-invasive ventilation; High flow oxygen therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- weaning group (Other): Patients included in the study will not be randomized individually but will be managed either according to the standard of care of the service or according to the personalized strategy (according to the stepped wedge group of the center).
  Interventions: Procedure: weaning by early non-invasive ventilation and progressive high flow oxygen therapy

INTERVENTIONS:
Procedure: weaning by early non-invasive ventilation and progressive high flow oxygen therapy — Step 1 Clinical stability was confirmed:
  (1)Without organ failure;(2)Without sepsis;(3)Stable heart rate and blood pressure without use of vascular active drugs.
  Step2 Reduce the support parameters of the ventilator gradually. Step3 SBT when the ventilator mode is pressure support ventilation(PSV),P+PEEP≤16cmH2O for 2 hours.
  Step4
  ①Success of SBT: titrate based HFOT time-------connected with tracheostomy tube ,flow rate and FiO2 able to maintain oxygen saturation as assessed by pulse oximetry monitoring of at least 95%.HFOT was interrupted in cases of sighs or symptoms of distress such as oxygen desaturation, RR>30bpm, HR>130bpm,SBP>180mmHg or <90mmHg.The time was based HFOT time. When any of these conditions were present the patient was connected again to the ventilator with the same parameters before titration. The duration of SBT was increased progressively over the following day according to patient tolerance. Then gradually extending HFOT time daily according patient condition. Wh

SUMMARY:
The aim of our study was to assess the feasibility of an early NIV and progressive HFOT through tracheostomy tube weaning protocol implemented by tracheostomized patients with PMV referred to a specialized weaning unit of a rehabilitation hospital.

DETAILED DESCRIPTION:
The most common indications for tracheostomy are acute respiratory failure with demonstrate or expected prolonged duration of mechanical ventilation (MV),failure to wean from MV.MV is associated with several complications. Placement of a long-term airway (tracheostomy) is also associated with short and long term risks. As more patients with multiple co-morbidities undergo tracheostomy and develop difficulty with weaning, new innovative concepts are urgently needed for their management. Surprisingly, there is very little data dealing with tracheostomized patients in weaning from mechanical ventilation and subsequent tracheostomy tube decannulation.

PMV patients were not able to sustain completely unsupported breathing ,since their load/capacity balance was impaired. Spontaneous breathing trial is not suitable for PMV patients.

For these reasons, PMV patients are often transferred to specialized weaning units with multidisciplinary teams ,which offer advanced weaning protocols and physiotherapists. The role of non-invasive ventilation(NIV) in MV patients with tracheostomy tube to facilitate both weaning off from the ventilator and removal of the tracheostomy tube has a solid physiological rationale, but most clinical evidence is derived from limited observational studies. And mainly focus on patients with chronic obstructive pulmonary disease(COPD) .Besides most NIV delivered through the facial interface while the tracheostomy tube is capped. This was difficult to tolerate for patients with poor lung function and upper airway obstruction. Then delayed NIV transfer. High flow oxygen therapy(HFOT)allows a more accurate FiO2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* After tracheotomy;
* Patients who met the definition of long-term mechanical ventilation (requiring invasive mechanical ventilation for more than 6 hours per day for more than 21 consecutive days);
* willing to participate in this study and signed the informed consent.

Exclusion Criteria:

* The expected survival time less than 3 months;
* Participated in another clinical study related to weaning;
* death or discharge within 2 weeks after referral;
* Unable to cooperate with the study for any reason or considered not suitable for inclusion in the trial by the investigators;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
weaning success | through study completion, an average of 100 days

SECONDARY OUTCOMES:
mechanical ventilation days | 120 days
  the duration of mechanical ventilation
weaning duration | through study completion, an average of 120 days
Length of stay | 6 months
1 year survival | 1 year
Rate of extubation | through study completion, an average of 100 days
Discharge destination | 12 months
  At hospital discharge, did the patient return Home or were they discharged to a post-acute care Rehab Facility
Mortality rate in hospital | 12 months
Re-hospitalization rate within 1 year | 12 months
Length of stay at HDU | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ge, Principal Investigator — Study Principal Investigator; Jingyi Ge, Principal Investigator — Beijing Rehabilitation Hospital of Capital Medical University
Locations (1):
- Beijing Rehabilitation Hospital of Capital Medical University, Beijing, China